## Screening of Patients With Suspected Heart Rhythm Disorder on Primary Health Care Level With the Use of Personal Digital ECG Sensor



26. 06. 2016 Staša Vodicka, MD

Health care center Murska Sobota

Grajska ulica 24, 9000 Murska Sobota

Slovenia

## PROJECT ECG SENSOR

Ambulanta Staša Vodička, dr. med., spec. druž. med. Zdravstveni dom Murska Sobota Grajska ulica 24, Murska Sobota

## Personal electrocardiogram - PCARD

## CONSENT for test use

You have agreed to test a small electrocardiogram (ECG) sensor on your own. The device measures the ECG, and the signal is wirelessly transmitted to the mobile phone where the MobEcg application runs. The ECG signal is visible on the phone screen, while the data is entered into the file, which allows for a later detailed analysis.

The device is in a test form and is not protected against water intrusion. It is, therefore, necessary to remove it before the shower. The battery on the device is filled with a special charger. The ECG on the body is installed with two self-adhesive electrodes in the appropriate chest position where it is not disturbing for you. At the same time, the ECG signal is good and contains all electrocardiographic waves (P, QRS and T). If your device is bothering you, remove it. Later, you can reinstall it to continue the measurement. The handling of the device will be presented in more detail before surrender.

The purpose of the test is for you to get familiar with the new possibility of monitoring the ECG. For us, your impressions and your ideas about the gadget are essential. After completing the test, we will analyze the recorded ECG. By signing, you acknowledge that you have received the device and will return it after a certain period.

By signing, you also acknowledge that you are aware of the operation of the device and its handling and to allow analysis of ECG measurements. In any scientific publication of the results of the studies, only your age and gender will be given. All other personal data will be erased.

This consensus exists in duplicate. The Volunteer receives one copy, and the other is the person who presented and surrendered the device.

| Name of volunteer: | Gender: Age: |
|---------------------------|----------------------------|
| Address: | |
| Device Pickup Date: | |
| Volunteer Signature: | _ |
| Device Label: | Date to return the device: |
| Date of Return of device: | Volunteer Signature: |

